CLINICAL TRIAL: NCT00692419
Title: Pain, Sexual Dysfunction and Depression in Hemodialysis Patients
Brief Title: Pain, Sexual Dysfunction, and Depression in Hemodialysis Patients
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Dialysis Clinic, Inc. (Industry); Liberty Dialysis, LLC (Other); DaVita, Inc. (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 07-190
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-09

CONDITIONS: End Stage Renal Disease; Sexual Dysfunction, Physiological; Pain; Depression
Keywords: pain; sexual dysfunction; depression; symptoms
MeSH Terms: conditions — Kidney Failure, Chronic; Sexual Dysfunction, Physiological; Pain; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symptom management nurse intervention (Experimental): This arm of the study will have a symptom management nurse facilitate the management of pain, sexual dysfunction and depression. The nurse will work with the patient's renal provider to implement appropriate symptom alleviating treatment. The intervention is patient specific and entirely dependent on the treatment recommendation made by the symptom management nurse.
  Interventions: Behavioral: Symptom management nurse intervention
- Feedback intervention (Active Comparator): This arm of the study will have pain, sexual dysfunction and depression assessed monthly with feedback given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider. The intervention on symptoms is at the discretion of the renal provider. The interventions implemented were patient specific and consisted of therapies the patient's renal provider decided to implement.
  Interventions: Behavioral: Feedback intervention

INTERVENTIONS:
Behavioral: Symptom management nurse intervention — A symptom management nurse will facilitate the management of pain, sexual dysfunction and depression in patients enrolled in one arm of the study
  Arms: Symptom management nurse intervention
Behavioral: Feedback intervention — Pain, sexual dysfunction and depression will be assessed monthly and feedback will be given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider
  Arms: Feedback intervention

SUMMARY:
This study is seeking to identify the most effective strategy to manage pain, sexual dysfunction, and depression in patients receiving chronic hemodialysis therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

There are currently over 500,000 individuals with end-stage renal disease (ESRD) in the United States, and more than 100,000 new patients develop this condition annually. Recent estimates suggest that more than 35,000 veterans currently receive chronic hemodialysis. Although life-sustaining, hemodialysis is associated with substantial morbidity and mortality. Numerous studies have sought to identify interventions that reduce the mortality of patients dependent on hemodialysis, yet recent clinical trials of dialysis dose, dialysis membrane, and lipid lowering therapy have failed to demonstrate survival benefits. With the recognition that providers have limited means beyond renal transplantation to prolong the lives of patients on hemodialysis, investigators are beginning to refocus their research efforts on identifying interventions to improve patients' quality of life, which is substantially impaired in this population. Several major factors that contribute to poor quality of life have been identified, including the large burden of physical and emotional symptoms in this patient population.

Of the many symptoms that affect patients on hemodialysis, pain, sexual dysfunction, and depression are among the most prevalent, severe, and highly correlated with impaired quality of life. These observations are particularly noteworthy with recent data documenting the safety and efficacy of pharmacologic therapy for these symptoms. Nonetheless, preliminary studies suggest that even when severe, these symptoms are untreated or under-treated in patients on hemodialysis. The reasons for the sub-optimal treatment have not been clearly elucidated, but the investigators research demonstrated that renal providers are largely unaware of the presence and severity of pain, sexual dysfunction, and depression in their hemodialysis patients. Although increasing provider awareness of these symptoms would seem to be important for the provision of therapy, it is not clear that simply informing clinicians would be sufficient to improve treatment.

The broad objective of this 3-year project is to determine the most effective strategy for the management of pain, sexual dysfunction, and depression in patients on chronic hemodialysis. The investigators postulate that merely informing renal providers of patients' pain, sexual dysfunction, and depression and providing them with evidence-based treatment algorithms will not significantly improve the management of these symptoms. Rather, optimal symptom management will require assessment and treatment of these symptoms by a dedicated renal symptom management nurse. In a randomized clinical trial of not more than 350 patients receiving hemodialysis at 9 dialysis units, the investigators will compare two symptom management strategies: (a) providing feedback on patients' symptoms to renal providers along with evidence-based algorithms for their treatment and; (b) using a renal symptom management nurse to identify and facilitate treatment of these symptoms. This study involves the nurse and the research assistant bringing treatment plans and algorithms to the attention of the renal providers and does not involve any treatment by the research assistant and nurse themselves. By determining the most effective approach to the management of overall pain, sexual dysfunction, and depression, the investigators hope to introduce a patient-centered management approach to improve the quality of life of patients receiving chronic hemodialysis.

METHODS: Overview of Study Design The investigators have proposed a randomized, clinical trial to compare two strategies for the treatment of pain, sexual dysfunction, and depression in patients on chronic hemodialysis. The investigators have recruited 315 patients from nine local VA and non-VA dialysis units.

After enrollment, baseline data was collected from 289 patients, and an observation period of at least 2 months but not longer than 12 months ensued. Pain, sexual dysfunction, and depression were assessed monthly during this observation period, which allowed us to establish the stability of symptoms in study patients and obtain a valid estimate of the impact of the investigators interventions on these domains. Additionally, quality of life, overall symptom burden and satisfaction with care was assessed every 3 months. The investigators assessment of sexual function focused on ED in men, and decreased libido, arousal, dyspareunia, and satisfaction in women. The investigators also conducted monthly assessments of patients' attendance at dialysis, compliance with treatment duration, emergency room visits, and hospitalizations.

After the observational phase, the investigators launched a 12-month intervention phase to compare two interventions. During this phase, the investigators continue these same assessments of pain, sexual dysfunction, depression, quality of life, overall symptom burden and satisfaction with care. The investigators continue to track attendance and compliance with dialysis, emergency room visits, and hospitalizations on a monthly basis. Patients are randomized into one of two study arms by day of dialysis treatment (Monday, Wednesday, and Friday versus Tuesday, Thursday, and Saturday). Sites that only treat patients on a Monday/Wednesday/Friday dialysis schedule are randomized by the time of the dialysis shift within the day, patients on the a.m. shift are randomized to one arm of the study and those on the p.m. shift to the other. One group is randomized to a "feedback intervention" in which renal providers will receive data on the presence and severity of patients' pain, sexual dysfunction, and depression along with algorithms for the treatment of these symptoms (For sexual dysfunction, providers will receive a treatment algorithm for ED and a recommendation to refer women with this symptom for gynecologic care). Treatment decisions will be left at the discretion of the provider(s). The other group has a renal symptom management nurse assess and facilitate the treatment of pain, sexual dysfunction, and depression (management intervention).In this arm, treatment of sexual dysfunction in men will focus on ED, while the symptom management nurse will facilitate referral of women with sexual dysfunction for gynecological care given the lack of pharmacologic therapy.

Study Status: Intervention Phase is completed, analysis is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Our target population is male and female hemodialysis patients age 18 years or greater who are English speakers.

Exclusion Criteria:

* We will exclude children because they comprise a minority of the dialysis population and their enrollment would require an adult decision maker's consent.
* We will exclude patients who are significantly cognitively impaired and hence, unable to comprehend study surveys.
* Cognitive function will be assessed at baseline using the mini-Cog, a validated measure of cognitive capacity that we have used previously, and patients with scores <3 will be excluded.
* Based on our prior studies, we estimate that approximately 5% of patients will be excluded based on this criterion.
* Similarly, non-English speakers will be excluded.
* Finally, patients undergoing active work-up for living donor kidney transplant, and/or considering transfer to peritoneal dialysis will be excluded as they are less likely to remain on hemodialysis for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Weisbord, MD MSc, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Weisbord SD, Shields AM, Mor MK, Sevick MA, Homer M, Peternel J, Porter P, Rollman BL, Palevsky PM, Arnold RM, Fine MJ. Methodology of a randomized clinical trial of symptom management strategies in patients receiving chronic hemodialysis: the SMILE study. Contemp Clin Trials. 2010 Sep;31(5):491-7. doi: 10.1016/j.cct.2010.06.005. Epub 2010 Jul 1. PMID 20601163
- [Result] Weisbord SD. Sexual dysfunction and quality of life in patients on maintenance dialysis. Semin Dial. 2013 May-Jun;26(3):278-80. doi: 10.1111/sdi.12068. Epub 2013 Mar 5. No abstract available. PMID 23458106
- [Result] Green JA, Mor MK, Shields AM, Sevick MA, Arnold RM, Palevsky PM, Fine MJ, Weisbord SD. Associations of health literacy with dialysis adherence and health resource utilization in patients receiving maintenance hemodialysis. Am J Kidney Dis. 2013 Jul;62(1):73-80. doi: 10.1053/j.ajkd.2012.12.014. Epub 2013 Jan 24. PMID 23352380
- [Result] Mor MK, Sevick MA, Shields AM, Green JA, Palevsky PM, Arnold RM, Fine MJ, Weisbord SD. Sexual function, activity, and satisfaction among women receiving maintenance hemodialysis. Clin J Am Soc Nephrol. 2014 Jan;9(1):128-34. doi: 10.2215/CJN.05470513. Epub 2013 Dec 19. PMID 24357510
- [Result] Weisbord SD, Mor MK, Sevick MA, Shields AM, Rollman BL, Palevsky PM, Arnold RM, Green JA, Fine MJ. Associations of depressive symptoms and pain with dialysis adherence, health resource utilization, and mortality in patients receiving chronic hemodialysis. Clin J Am Soc Nephrol. 2014 Sep 5;9(9):1594-602. doi: 10.2215/CJN.00220114. Epub 2014 Jul 31. PMID 25081360
- [Result] Green JA, Mor MK, Shields AM, Sevik MA, Palevsky PM, Fine MJ, Arnold RM, Weisbord SD. Renal provider perceptions and practice patterns regarding the management of pain, sexual dysfunction, and depression in hemodialysis patients. J Palliat Med. 2012 Feb;15(2):163-7. doi: 10.1089/jpm.2011.0284. PMID 22339326
- [Result] Weisbord SD. Female sexual dysfunction in ESRD: an underappreciated epidemic? Clin J Am Soc Nephrol. 2012 Jun;7(6):881-3. doi: 10.2215/CJN.03870412. Epub 2012 May 10. No abstract available. PMID 22580787
- [Result] Weisbord SD, Mor MK, Green JA, Sevick MA, Shields AM, Zhao X, Rollman BL, Palevsky PM, Arnold RM, Fine MJ. Comparison of symptom management strategies for pain, erectile dysfunction, and depression in patients receiving chronic hemodialysis: a cluster randomized effectiveness trial. Clin J Am Soc Nephrol. 2013 Jan;8(1):90-9. doi: 10.2215/CJN.04450512. Epub 2012 Sep 27. PMID 23024159
- [Result] Green JA, Mor MK, Shields AM, Sevick MA, Palevsky PM, Fine MJ, Arnold RM, Weisbord SD. Prevalence and demographic and clinical associations of health literacy in patients on maintenance hemodialysis. Clin J Am Soc Nephrol. 2011 Jun;6(6):1354-60. doi: 10.2215/CJN.09761110. Epub 2011 May 5. PMID 21551025
- [Result] Belayev LY, Mor MK, Sevick MA, Shields AM, Rollman BL, Palevsky PM, Arnold RM, Fine MJ, Weisbord SD. Longitudinal associations of depressive symptoms and pain with quality of life in patients receiving chronic hemodialysis. Hemodial Int. 2015 Apr;19(2):216-24. doi: 10.1111/hdi.12247. Epub 2014 Nov 18. PMID 25403142
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: the number of patients recruited into the study beginning at the time of the observation phase (315) differs from the number of patients who continued in the study and were included in the intervention phase of the study (220)
Groups:
- Arm 1: This arm of the study will have a symptom management nurse facilitate the management of pain, sexual dysfunction and depression
  Renal Symptom Management Nurse Practitioner Intervention: A symptom management nurse will facilitate the management of pain, sexual dysfunction and depression in patients enrolled in one arm of the study
- Arm 2: This arm of the study will have pain, sexual dysfunction and depression assessed monthly with feedback given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider
  Feedback of Symptoms Intervention: Pain, sexual dysfunction and depression will be assessed monthly and feedback will be given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 100 | 120
Completed | 84 | 102
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Symptom Management Intervention: This arm of the study will have a symptom management nurse facilitate the management of pain, sexual dysfunction and depression
  Renal Symptom Management Nurse Practitioner Intervention: A symptom management nurse will facilitate the management of pain, sexual dysfunction and depression in patients enrolled in one arm of the study
- Feedback Intervention: This arm of the study will have pain, sexual dysfunction and depression assessed monthly with feedback given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider
  Feedback of Symptoms Intervention: Pain, sexual dysfunction and depression will be assessed monthly and feedback will be given to renal providers on the presence and severity of these symptoms. Treatment will be left at the discretion of the renal provider
- Total: Total of all reporting groups
Arm/Group | Symptom Management Intervention | Feedback Intervention | Total
Number analyzed (Participants) | 100 | 120 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.3) | 63.9 (12.0) | 63.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 55 | 99
  Male | 56 | 65 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain, Sexual Dysfunction, and Depression Symptoms
Description: The primary outcome of this study is the change in symptom scores during the intervention phase of the study
Time Frame: 12 months
Population: change in pain score during intervention period. In adjusted models, we used mixed effects linear regression to compare changes in symptom scores between the two study arms over the duration of the intervention, and to compare symptom scores among individual patients across the observation and intervention phases.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Management Arm Change in Pain Score: Management arm change in pain score of the Short Form McGill Pain Questionnaire (SF-MPQ) during the intervention. The SF-MPQ includes 15 pain descriptors that are rated from 0 (no pain) to 3 (severe pain), with a summary score of 0-45. Higher scores represent more pain.
- Feedback Group - Change in Pain Score: Feedback group - change in pain score of the Short Form McGill Pain Questionnaire (SF-MPQ) during the intervention. The SF-MPQ includes 15 pain descriptors that are rated from 0 (no pain) to 3 (severe pain), with a summary score of 0-45. Higher scores represent more pain.
- Management Group - Change in ED Score: Management group - change in ED score on the Sexual Health Inventory for Men (SHIM) questionnaire during the intervention. We scored the SHIM from 5-25 with lower scores denoting more severe ED. We considered patients with SHIM scores <22 to have ED.
- Feedback Group - Change in ED Score: Feedback group - change in ED score on the Sexual Health Inventory for Men (SHIM) questionnaire during the intervention. We scored the SHIM from 5-25 with lower scores denoting more severe ED. We considered patients with SHIM scores <22 to have ED.
- Management Group - Change in Depression Score: Management group - change in depression score on the Patient Health Questionnaire 9 (PHQ-9) during the intervention. The PHQ-9 is scored from 1 to 27, with higher scores denoting more severe depression. We considered patients with PHQ-9 scores ≥10 to have depression.
- Feedback Arm Change in Depression Score: Feedback arm change in depression score on the Patient Health Questionnaire 9 (PHQ-9) during the intervention. The PHQ-9 is scored from 1 to 27, with higher scores denoting more severe depression. We considered patients with PHQ-9 scores ≥10 to have depression.
Arm/Group | Management Arm Change in Pain Score | Feedback Group - Change in Pain Score | Management Group - Change in ED Score | Feedback Group - Change in ED Score | Management Group - Change in Depression Score | Feedback Arm Change in Depression Score
Number analyzed (Participants) | 100 | 120 | 100 | 120 | 100 | 120
units on a scale | -3.12 (0.54) | -3.7 (0.51) | 0.62 (0.34) | 0.71 (0.32) | -1.99 (0.54) | -2.29 (0.49)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 19/100 | 15/120
Other Adverse Events (participants affected / at risk) | 2/100 | 1/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=100) | Arm 2 (N=120)
death (General disorders) | 19 (19) | 15 (15) — These are the # of deaths. However, none of these deaths were thought related to study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=100) | Arm 2 (N=120)
medication side effect (Nervous system disorders) | 2 (100) | 1 (120) — the event was characterized as medication side effect

LIMITATIONS AND CAVEATS:
Individual providers were overseeing the care of patients from both study arms. The sample size was relatively small. Single geographic area. No control arm. Symptoms assessed during dialysis. No formal assessment of treatment compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes